CLINICAL TRIAL: NCT04537468
Title: Development of a Method to Measure mRNA Levels From the Skin of Patients With Psoriasis and Patients With Atopic Dermatitis Using Tape Strippings
Brief Title: Development of a Method to Measure mRNA Levels in Skin Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Inno-5001
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy; Atopic Dermatitis Eczema; Psoriasis
Keywords: Skin squames; Tape stripping; Skin biopsy
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: The study consisted of 3 sequential groups:
  1. Collection of skin squames by scraping.
  2. Collection of tape strip samples.
  3. Collection of tape strip samples and skin biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin sample collection (Other): Skin sample collection for gene expression analyses.
  Interventions: Other: Skin squame collection; Other: Tape strip collection; Other: Tape strip and skin biopsy collection

INTERVENTIONS:
Other: Skin squame collection — Subjects underwent skin squame collection by scraping. The investigator gently scraped the surface of a lesional skin area for patients with psoriasis, and of a non-lesional skin area for healthy volunteers to collect superficial cells. These samples were analyzed by gene expression analyses.
Other: Tape strip collection — The first subjects had up to 35 tape strips from a maximum of 4 areas (4 X 35 strippings) on the trunk or limbs (excluding the genital area). Patients with atopic dermatitis or psoriasis had tape stripping performed on lesional skin areas and the control subjects had tape stripping performed on nonlesional skin areas. The next subjects were used to determine the optimal number of tape strips required to obtain a good signal by gene expression analyses.
Other: Tape strip and skin biopsy collection — Subjects had tape stripping on up to 3 different skin areas (2 areas on lesional skin and one area of nonlesional skin for patients with atopic dermatitis or psoriasis, and 2 areas of healthy skin for control subjects) using the optimal number of tape strips, as determined in the previous part. One 4-mm skin biopsy on a tape stripped area plus one 4-mm biopsy on non-tape-stripped skin (2 biopsies per subject) were also collected.

SUMMARY:
The purpose of this study was to develop a non-invasive method to measure mRNA levels using tape stripping on the skin of patients with psoriasis and patients with atopic dermatitis.

DETAILED DESCRIPTION:
Three sequential groups of subjects were recruited in this study for: 1) skin squame collection; 2) tape strip collection; and 3) tape strip and skin biopsy collection in the aim of identifying the most optimal method for measuring the mRNA levels of skin biomarkers in tape strip samples.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, aged 18 years or older at the time of consent.
* Female subjects of childbearing potential had a negative urine pregnancy test at the screening visit.
* Subjects had to be able and willing to provide written informed consent and comply with the requirements of the study protocol. Consent was obtained prior to any study-related procedures.

  *Special inclusion criteria for volunteers with atopic dermatitis or psoriasis:
* Patient had a history of atopic dermatitis or psoriasis.
* Patient with psoriasis had a Physician's Global Assessment (PGA) score of ≥2 at Day 0.
* Patients with atopic dermatitis had an Investigator's Global Assessment (IGA) score of ≥2 at Day 0.

Exclusion Criteria:

* Female subject was pregnant or breastfeeding.
* Subject was participating in a clinical trial with an experimental drug or device or had participated in a clinical trial with an experimental drug or device within the last 4 weeks of the collection day (Day 0).
* Subject was known to have hepatitis B or hepatitis C viral infection.
* Subject was known to have immune deficiency or was immunocompromised.
* Subject had used systemic medication, medical devices, UVB or PUVA therapy or natural health products to treat atopic dermatitis or psoriasis on the areas to be biopsied or tape stripped within 4 weeks of the collection day (Day 0).
* Subject had used oral, intravenous steroids, or immunosuppressive medication within 4 weeks of the collection day (Day 0). Subject had used intramuscular or intra-lesional or intra-articular steroids or immunosuppressive medication on the areas to be biopsied or tape stripped within 4 weeks of the collection day (Day 0).
* Subject had used a biologic within 12 weeks or 5 half-lives of the collection day (Day 0), whichever was longer.
* Subject had used topical medication, natural health products or medical devices to treat atopic dermatitis or psoriasis on the areas to be tape stripped or biopsied within 2 weeks of the collection day (Day 0).

  *Only for subjects who underwent skin biopsy:
* Subject had a known hypersensitivity/allergy to lidocaine.
* Subject had a history of hypertrophic scarring or keloid formation in scars or suture sites.
* Subject was taking anti-coagulant medication (e.g. heparin, low molecular weight [LMW]-heparin, warfarin, anti-platelets [nonsteroidal anti-inflammatory drugs (NSAIDs) and low-dose aspirin (equal or lower than 81 mg) were not considered anti-platelets]) or had a contraindication to skin biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Expression of skin biomarkers | Day 0
  Gene expression of epidermal cytokines and chemokines.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research, Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He H, Bissonnette R, Wu J, Diaz A, Saint-Cyr Proulx E, Maari C, Jack C, Louis M, Estrada Y, Krueger JG, Zhang N, Pavel AB, Guttman-Yassky E. Tape strips detect distinct immune and barrier profiles in atopic dermatitis and psoriasis. J Allergy Clin Immunol. 2021 Jan;147(1):199-212. doi: 10.1016/j.jaci.2020.05.048. Epub 2020 Jul 21. PMID 32709423